CLINICAL TRIAL: NCT05381584
Title: Balloon Vaginoplasty; Fully Monitored Entry Versus Fractionated Intraumbilical Microports for Treatment of Vaginal-aplasia; A Quasi Randomized Controlled Trial
Brief Title: Balloon Vaginoplasty for Treatment of Vaginal-aplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alshimaa Hassan Hosney Eeraqi, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: vagioplasty in vaginal aplasia
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Vaginal Abnormality
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fractionated intraumbilical microports group (Active Comparator): two 4-5-mm micro ports will be done intra umbilically; a 4-mm scope is inserted through one of them, followed by a 4-mm catheter inserter through the second intra umbilical port.
  Interventions: Procedure: laparoscopy
- fully monitored entry group (Experimental): only one 4mm intra umbilical port will be done and a second port at a point of lies 8 cm from midline and 5 cm above anterior superior iliac spine. After performing laparoscopic evaluation of the pelvis the telescope will be moved from the umbilical port to the ancillary port and the catheter loaded inserter will be introduced through the umbilical port its insertion will be fully monitored from the point of entry at the umbilicus until the pelvic floor.
  Interventions: Procedure: laparoscopy

INTERVENTIONS:
Procedure: laparoscopy — laparoscopy will be done under anesthesia for management for cases with blind vagina

SUMMARY:
Vaginal aplasia is a congenital anomaly characterized by congenital absence of the vagina with an incidence approximately 1:4,500-6,000. It carries an emotional, sexual, and social embarrassing effect on those women, The primary aim of treatment is creation of a neo vagina for restoration of the ability for vaginal intercourse. There are several techniques for neo vaginal construction with variable satisfaction rates. Most of these procedures are either invasive and technically demanding or require long duration in a very motivated patient

DETAILED DESCRIPTION:
Numerous surgical and nonsurgical procedures with varying degrees of success have been described for correction of the vaginal aplasia, but none have proved to be universally accepted.

Balloon vaginoplasty was first introduced in 2003 by El Saman et al for construction of a naturally lined neo vagina through a laparoscopic.

Technique hosts the triad of a perfect management modality; namely: simplicity, safety and success. The technique acts via mechanical expansion of the vaginal epithelium and underlying tissues at the pre-existing vaginal dimple Being a relatively new modality of management, it went through many refinements to make it much easier and feasible. The cornerstone of refinement always ran around the access to the peritoneal cavity. The latest of which was the fractionated intra umbilical micro ports which have the merits of totally hidden scar at the bottom the umbilicus consequently the best cosmetic outcomes. However, during its insertion process a troublesome partially unmonitored insertion was inevitably observed

ELIGIBILITY:
Inclusion Criteria:

* Married Females with vaginal aplasia scheduled for balloon vaginoplasty.

Exclusion Criteria:

* Females who refused to consent for participation in the study.
* Unstable marital relationship.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The Operative time | 1 hour
  duration of surgery will be calculated from start of laparoscopy